CLINICAL TRIAL: NCT00623688
Title: Effectiveness and Costs of Albuterol Delivered by MDI With Spacer Versus Nebulizer in Children Hospitalized With Moderate and Severe Asthma Exacerbations
Brief Title: Effectiveness and Cost Study Comparing Two Ways to Deliver Albuterol for the Treatment of Asthma in the Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akron Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 070908
Record Dates: First submitted 2008-02-06; First posted 2008-02-26 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Status Asthmaticus
Keywords: Metered Dose Inhalers; Nebulizers; Randomized Controlled Trial
MeSH Terms: conditions — Status Asthmaticus | interventions — Metered Dose Inhalers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Subjects receive active medication (albuterol) delivered by a Proair metered dose inhaler used with an Opti-chamber and placebo (normal saline solution) by nebulizer aerosol.
  Interventions: Device: Metered Dose Inhaler & Optichamber Advantage Valve Holding Chamber (VHC)
- 2 (Active Comparator): Subjects receive active medication (albuterol) delivered by nebulizer and placebo (no medicine) delivered by a demonstrator Placebo metered dose inhaler demonstrator.
  Interventions: Device: Airlife Sidestream High Efficiency Nebulizer

INTERVENTIONS:
Device: Metered Dose Inhaler & Optichamber Advantage Valve Holding Chamber (VHC) — Albuterol is delivered by metered dose inhaler with valved holding chamber. For children less than 6 years of age, a mask is also used.
  Arms: 1
Device: Airlife Sidestream High Efficiency Nebulizer — Albuterol is delivered as a mist mixed with normal saline using a nebulizer machine and face mask or mouth piece.
  Arms: 2

SUMMARY:
This study will be conducted as a randomized, double blinded, controlled trial. The control group will receive albuterol delivered by a nebulizer along with placebo treatments delivered by a metered dose inhaler (MDI) with a spacer +/- mask. The experimental group will receive albuterol delivered by MDI with spacer +/- mask along with placebo treatments given by a nebulizer. Parents, participants, study personnel, nursing staff, and respiratory therapists will not know the treatment assignments of participants. The primary outcome will be changes over time in an asthma severity score, the Clinical Asthma Score (CAS) (Parkin et al. 1996). The secondary outcomes will be total number of albuterol treatments received in the hospital, time it take to give treatments, time till subjects' albuterol treatments are given at four hour intervals, and the costs of the two types of treatments. The study hypothesis is that albuterol delivered by metered dose inhaler with spacer is non-inferior to albuterol delivered by nebulizer in the treatment of children hospitalized with moderate to severe asthma exacerbations.

DETAILED DESCRIPTION:
Studies looking at the use of beta-2-agonists given by MDIs with a spacer and mask in children greater than 2 years have described fewer side effects than when the same medications are given as nebulizers. Patients have less tachycardia, vomiting, and oxygen desaturation (Kerem et al. 1993, Chou, Cunningham and Crain 1995, Lin and Hsieh 1995, Pendergast et al. 1989, Fuglsang and Pedersen 1986).

In the emergency department setting, Rubilar et. al found that albuterol delivered by MDI with spacer and mask had equal efficacy to albuterol delivered by a nebulizer in treating acute wheezing in children less than 2 years of age. (Rubilar, Castro-Rodriguez and Girardi 2000) Chou et. al found that in children greater than 2 years old with acute asthma exacerbations, MDIs had the same efficacy as nebulizers but with a shorter delivery time and fewer side effects.(Chou et al. 1995)

All children who meet criteria to be participants in the study will be approached for possible study enrollment in the ED. No outside recruiting will be done. Once consent has been obtained and patients are enrolled, they will be randomized to either albuterol by MDI with placebo nebulizer treatments or albuterol by nebulizer with placebo MDI treatments. Subjects will be randomized to one of the two treatment arms in a 1:1 randomization process. This will be done using a prepared assignment log developed using a random number generator.

Children in the control arm will receive albuterol via nebulizer and placebo by MDI with spacer +/- mask. Children in the experimental arm will receive albuterol by MDI and placebo by nebulizer.

All MDI treatments will be given with a spacer +/- mask. Subjects will receive 6 puffs if they are < 30 kg and 10 puffs if they are > 30 kg. If they are in the control group, puffs will be placebo. If they are in the experimental group, puffs will be albuterol (90 micrograms per puff).

For the nebulizer treatments, patients in the control group will receive 2.5 mg albuterol (if <30 kg) or 5 mg of albuterol (if 30 kg or greater) in 3 ml of normal saline. Patients in the experimental group will receive nebulizer treatments as 3 ml of normal saline. Nebulized treatments will be delivered with room air unless the subjects are on oxygen.

All study medication will be administered by clinical nursing staff or respiratory therapists. The frequency at which albuterol is given will be determined by the subject's primary medical team. For all subjects, MDI treatments will be given first followed by nebulizer treatments.

Nursing staff will record a Clinical Asthma Score (CAS) (Parkin et. al 1996) on admission and every 4 hours during hospitalization up to 72 hours or discharge (whichever comes first). Nursing staff will also record the total number of albuterol treatments given and the time required to give each treatment. Patients' total length of stay will be calculated. A cost analysis will be done to determine if there are any differences in the costs to the hospital of the two delivery devices. This analysis will include the costs of the albuterol and delivery devices and the labor costs related to nursing or respiratory therapists' time to administer the medications. Information on subjects' baseline level of asthma severity will also be collected at the beginning of the study.

All study patients will be given prednisolone, prednisone or solumedrol at a dose of 1 mg/kg/dose twice a day for a total of 5 days. The length of steroid treatment can be extended beyond 5 days if felt to be clinically indicated by the subject's attending physician.

Controller medications such as long acting beta-2-agonists, inhaled corticosteroids, and leukotriene inhibitors will be given at the discretion of the subject's in patient attending. All controller medications used before and during hospitalization will be recorded as part of the study data.

ELIGIBILITY:
Inclusion Criteria:

* Children 1 to 18 years of age with a known history of asthma being admitted to Akron Children's Hospital general medical floor for the treatment of moderate to severe asthma exacerbations

Exclusion Criteria:

* Children who have a concurrent pneumonia or bronchiolitis (diagnosed clinically or by chest x-ray)
* Have a diagnosis of chronic lung disease (ex. cystic fibrosis, bronchopulmonary dysplasia, chronic aspiration)
* Have cyanotic congenital heart disease, a congenital anomaly of the respiratory tract, or who are tracheostomy or ventilator dependent.
* Children who are determined by the Emergency Department (ED) or general pediatrics service to need ICU level care on admission will also be excluded.
* Children will also be excluded if their legal guardian does not speak English as all consent forms will be written and reviewed with guardians in English.
* Children will also be excluded if their legal guardians disagree on consent to participate, or if a child 9 years or older and their legal guardians disagree on study participation.

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2008-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Change in Clinical Asthma Severity score over time | 72 hours

SECONDARY OUTCOMES:
Time to discharge | Total time in the hospital
Time to when are able to go 4 hours between albuterol treatments | Time in hospital
Cost of delivering albuterol by MDI versus nebulizer | Time in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly A Spoonhower, M.D., Principal Investigator — Akron Children's Hospital
Locations (1):
- Akron Children's Hospital, Akron, Ohio, United States

REFERENCES:
- [Background] Chou KJ, Cunningham SJ, Crain EF. Metered-dose inhalers with spacers vs nebulizers for pediatric asthma. Arch Pediatr Adolesc Med. 1995 Feb;149(2):201-5. doi: 10.1001/archpedi.1995.02170140083015. PMID 7849885
- [Background] Fuglsang G, Pedersen S. Comparison of Nebuhaler and nebulizer treatment of acute severe asthma in children. Eur J Respir Dis. 1986 Aug;69(2):109-13. PMID 3758239
- [Background] Kerem E, Levison H, Schuh S, O'Brodovich H, Reisman J, Bentur L, Canny GJ. Efficacy of albuterol administered by nebulizer versus spacer device in children with acute asthma. J Pediatr. 1993 Aug;123(2):313-7. doi: 10.1016/s0022-3476(05)81710-x. PMID 8345434
- [Background] Lin YZ, Hsieh KH. Metered dose inhaler and nebuliser in acute asthma. Arch Dis Child. 1995 Mar;72(3):214-8. doi: 10.1136/adc.72.3.214. PMID 7741566
- [Background] Parkin PC, Macarthur C, Saunders NR, Diamond SA, Winders PM. Development of a clinical asthma score for use in hospitalized children between 1 and 5 years of age. J Clin Epidemiol. 1996 Aug;49(8):821-5. doi: 10.1016/0895-4356(96)00027-3. PMID 8699199
- [Background] Pendergast J, Hopkins J, Timms B, Van Asperen PP. Comparative efficacy of terbutaline administered by Nebuhaler and by nebulizer in young children with acute asthma. Med J Aust. 1989 Oct 2;151(7):406-8. doi: 10.5694/j.1326-5377.1989.tb101224.x. PMID 2677624
- [Background] Rubilar L, Castro-Rodriguez JA, Girardi G. Randomized trial of salbutamol via metered-dose inhaler with spacer versus nebulizer for acute wheezing in children less than 2 years of age. Pediatr Pulmonol. 2000 Apr;29(4):264-9. doi: 10.1002/(sici)1099-0496(200004)29:43.0.co;2-s. PMID 10738013